CLINICAL TRIAL: NCT03208322
Title: Early Post-marketing Study of Daclatasvir (Daklinza®) + Asunaprevir (Sunvepra®) in the Treatment of Chronic Hepatitis C (CHC) in Adults
Status: Withdrawn | Type: Observational
Why Stopped: There was a change in the strategy to complete the RMP with HA.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI447-121
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- DCV + ASV at a sentinel site: patients with chronic hepatitis C (CHC) who are being given at least 1 dose of daclatasvir (DCV) and asunaprevir (ASV) for the treatment and cure of CHC at the sentinel sites for the National Pharmacovigilance Center (CNFV) in Mexico.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
The primary objective of the study is to determine the number of adverse events (AEs) reported by chronic hepatitis C (CHC) patients receiving at least 1 dose of daclatasvir (DCV) and asunaprevir (ASV) at the 2 sentinel sites and that have been reported through the Mexican Health Authority's AE surveillance system during a specified 24-month study period. The secondary objective is to describe AEs reported by CHC patients receiving treatment with DCV and ASV treated by doctors at participating sentinel sites for the National Pharmacovigilance Center (CNFV) in Mexico during a specified 24-month study period.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb (BMS) Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* at least 18 years of age with CHC, GT-1
* treatment-naïve and treatment-experienced (null or partial) responders
* intolerant to interferon (IFN)
* with or without cirrhosis

Exclusion Criteria:

* patients who received DCV and ASV as part of a clinical trial
* patients who received DCV and ASV for any indication other than that which is locally approved
* contraindications included in the approved Mexican prescribing information

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients receiving at least 1 dose of DCV and ASV at the selected sites during the specified 24 month study period. Included patients will be:
  * At least 18 years of age with CHC, Genotype(GT)-1
  * Treatment-naïve and treatment-experienced (null or partial) responders
  * Intolerant to interferon (IFN)
  * With or without cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
The number of adverse events (AEs) reported by patients treated with at least one dose of daclatasvir (DCV) and at least one dose of asunaprevir (ASV) and reported to the Health Authority (HA) during a specified period. | 24 months

SECONDARY OUTCOMES:
The adverse events (AEs) reported to the Health Authority (HA) during a specified period in table format identifying the report number, patient Identification number, and type of adverse event (AE). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Mexico (2):
  - Local Institution, Df, Mexico City
  - Local Institution, Magdalena de las Salinas, Mexico City

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm